CLINICAL TRIAL: NCT06333184
Title: Examining the Blood Sugar Response to Fruit Smoothie Consumption
Brief Title: Smoothies and Blood Sugars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, Professor of Nutrition and Metabolism, University of Bath
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 3085-4215
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Metabolic Disturbance
MeSH Terms: interventions — Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Control (Active Comparator): 50 g glucose (55 g dextrose powder accounting for hydration) plus 417 mL water
  Interventions: Other: Food
- Product (Experimental): 417 mL of commercially available "Mango & Passion fruit" fruit smoothie providing 50 g carbohydrate
  Interventions: Other: Food
- Whole (Experimental): Apples (51%), Mango (16%), Banana (16%), Orange (12%), Passionfruit (3%), Peach (2%), Lime (0.4%; recipe matched to PRODUCT) eaten as whole fruit with added water as needed to match volume.
  Interventions: Other: Food
- Blend (Experimental): Apples (51%), Mango (16%), Banana (16%), Orange (12%), Passionfruit (3%), Peach (2%), Lime (0.4%; recipe matched to PRODUCT) eaten as blended fruit with added water as needed to match volume.
  Interventions: Other: Food
- Slow (Experimental): 417 mL of commercially available "Mango and Passionfruit" fruit smoothie providing 50 g carbohydrate ingested slowly over 25-35 mins.
  Interventions: Other: Food
- Fibre (Experimental): 417 mL of commercially available "Mango and Passionfruit" fruit smoothie providing 50 g carbohydrate with 6 g of added inulin.
  Interventions: Other: Food
- Dose (Experimental): 250 mL of commercially available "Mango and Passionfruit" fruit smoothie providing 30 g carbohydrate.
  Interventions: Other: Food

INTERVENTIONS:
Other: Food — Fruit ingested in whole form or as either commercially available, or home-made smoothies

SUMMARY:
Glycaemic responses to fruit smoothies may depend on the food matrix (e.g., degree of processing and physical structure), ingestion rate, dose ingested and fibre content. Furthermore, the method of sampling could alter inferences. The aim of this project is to characterise how these factors affect the glycaemic response to a commercially available fruit smoothie. Participants will ingest 7 different test drinks in a randomised, crossover design with fingerstick capillary blood sampling alongside continuous glucose monitors. Test drinks will include a glucose reference (CONTROL), the commercial product matched for carbohydrate to CONTROL (PRODUCT), equivalent carbohydrate ingested as whole fruits (WHOLE), equivalent carbohydrate ingested as blended fruits (WHOLE), equivalent carbohydrate as the commercial product ingested slowly (SLOW), equivalent carbohydrate as the commercial product ingested with additional fibre (FIBRE), and the commercial product ingested in a dose typically bought (DOSE). These data will provide insight into how the food matrix and different patterns of ingestion can alter the glycaemic response to a fruit smoothie, and how the measurement method may alter interpretations.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* Body mass index 18-30 kg/m2

Exclusion Criteria:

* diagnosis of any form of diabetes
* intolerances or allergies to any of the study procedures (e.g. fructose/inulin intolerance)
* Fructose malabsorption
* Inborn errors of fructose metabolism (e.g. fructokinase deficiency, aldolase B deficiency, fructose-1,6-bisphosphatase deficiency)
* pregnant or lactating
* any condition that could introduce bias to the study (e.g. diagnoses of lipid disorders, including cardiovascular disease, or therapies that alter lipid or glucose metabolism, such as statins or niacin).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Glycaemic index of product with capillary vs CGM | 120 min
  The difference in glycaemic index [2-hour incremental area under the curve (mmol/L-1x120 min) for PRODUCT relative to CONTROL expressed as a percentage] in capillary blood samples versus continuous glucose monitors.

SECONDARY OUTCOMES:
Glycaemic index of all conditions with capillary vs CGM | 120 min
  The difference in glycaemic index [2-hour incremental area under the curve (mmol/L-1x120 min) for all other conditions (WHOLE, BLEND, SLOW, FIBRE, DOSE) relative to CONTROL expressed as a percentage] in capillary blood samples versus continuous glucose monitors.

OTHER OUTCOMES:
Condition-by-sampling interaction | 120 min
  The effect of condition-by-blood sampling (capillary vs continuous glucose monitor) interaction for the 2-hour incremental area under the curve for all conditions.
GI of products in capillary samples | 120 min
  Comparisons between conditions for the 2-hour incremental area under the curve relative to CONTROL using capillary blood glucose.
GI of products in continuous glucose monitors | 120 min
  Comparisons between conditions for the 2-hour incremental area under the curve relative to CONTROL using continuous glucose monitors.
Peak glucose capillary vs CGM | 120 min
  The condition-by-blood sampling interaction for the postprandial peak glucose concentrations (mmol/L)
Time to peak glucose capillary vs CGM | 120 min
  The condition-by-blood sampling interaction for the time to peak glucose concentrations (min)

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Health, University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available open access on the University of Bath Research Data Archive (RDA) at the point of publication in a peer-reviewed journal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: These will become available at the point of publication permanently.
URL: https://researchdata.bath.ac.uk/

REFERENCES:
- [Background] Gonzalez JT. Are all sugars equal? Role of the food source in physiological responses to sugars with an emphasis on fruit and fruit juice. Eur J Nutr. 2024 Aug;63(5):1435-1451. doi: 10.1007/s00394-024-03365-3. Epub 2024 Mar 16. PMID 38492022
- [Derived] Hutchins KM, Betts JA, Thompson D, Hengist A, Gonzalez JT. Continuous glucose monitor overestimates glycemia, with the magnitude of bias varying by postprandial test and individual - a randomized crossover trial. Am J Clin Nutr. 2025 May;121(5):1025-1034. doi: 10.1016/j.ajcnut.2025.02.024. Epub 2025 Feb 26. PMID 40021059